CLINICAL TRIAL: NCT00766766
Title: Reduction of Environmental Tobacco Smoke (ETS) Exposure In Pediatric Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: SMOKN5; 5R01CA085406 (NIH)
Record Dates: First submitted 2008-10-03; First posted 2008-10-06 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2013-09

CONDITIONS: Cancer
Keywords: Environmental Tobacco Exposure
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Experimental Intervention Group
  Interventions: Behavioral: Health Risk and Behavioral Skills Coaching Sessions; Behavioral: Telephone Coaching Sessions; Behavioral: Physician Feedback Letter
- 2 (No Intervention): Standard Care Control

INTERVENTIONS:
Behavioral: Health Risk and Behavioral Skills Coaching Sessions — Health Risk and Behavioral Skills Coaching Sessions
  Arms: 1
Behavioral: Telephone Coaching Sessions — Telephone Coaching Sessions
  Arms: 1
Behavioral: Physician Feedback Letter — Physician Feedback Letter
  Arms: 1

SUMMARY:
SMOKN5 is aimed at studying ways to reduce environmental tobacco smoke (ETS) for children who are being treated for cancer. The study includes St. Jude parents whose child lives with at least one adult smoker who exposes the child to ETS, also called "secondhand smoke." We are comparing two groups of parents to see which group results in lower ETS exposure levels for the child being treated with cancer. The first group will receive the standard information and advice usually given to parents about secondhand smoke. The second group will take part in a new program designed to reduce ETS. The primary objective of the study is to determine the efficacy of an environmental tobacco smoke intervention compared to the standard care control condition, as measured by parent report. Parents in each group answer questions about ETS exposure. We also collect urine samples from the child at specific time points throughout the study. The urine is tested to measure the amount of cotinine, a metabolite of nicotine. Measuring cotinine tells us how much nicotine from tobacco smoke the child has been exposed to. Children who are at least 10 years of age or older will also be asked to complete a set of questions pertaining to their tobacco use history and ETS exposure from others. This will occur at the same five time points in which the parent completes his/her portion. The study will last about 12 months for each participating family. Parents who take part in the study may learn how to lower their child's exposure to ETS, and this may, in turn, lower the child's chances of having ETS-related health problems.

DETAILED DESCRIPTION:
160 St. Jude families with a cancer patient who meets eligibility criteria will be enrolled on the study. Eligible St. Jude patients must be 17 years of age or younger at the time of enrollment. They must also be at least one month from initial diagnosis and in active treatment. The patient cannot currently be using tobacco, and he/she must live with at least one cigarette smoking adult who smokes in his/her presence. Both smoking and non-smoking parents are eligible to participate. The inclusion of non-smoking parents reflects the primary objective of the proposed study to reduce ETS exposure in the child's environment. We will evaluate the efficacy of an ETS intervention by using a randomized controlled trial design that incorporates an experimental intervention group (ETS) and a standard care control group (SCC). Parents in the SCC group will receive the standard advice with no additional intervention. The experimental group will participate in a three month, multi-component behavioral program focused on the reduction of the cancer patient's ETS exposure. The program will consist of three bi-weekly face-to-face coaching sessions followed by three bi-weekly telephone coaching sessions that will occur within the first three months following enrollment onto the study. Although telephone counseling sessions will be offered for parents who are not available in person, the face-to-face sessions are encouraged as much as possible. Parents in this group will receive physician feedback letters acknowledging their participation and progress at the start and end of the coaching phase, as well as, a follow-up telephone contact at five months. Self-report and biological measures will be obtained from all families during clinic visits at baseline and at three, six, nine, and twelve months. Reported ETS exposure and the child's urine cotinine levels will serve as the primary dependent variables. Other psychosocial and health outcomes will also be assessed. Children 10 years of age and older will complete a brief ETS exposure questionnaire that asks them to report on exposure in their environment. Parents in each group will be paid $10 for each set of study forms they answer. The total amount that a parent in the control group may receive is $50. Parents in the ETS intervention program will also receive $12.50 for each face-to-face and telephone coaching session in which they take part. The telephone follow-up call occurring at five months will not be compensated. The total amount that a parent in the ETS intervention group may receive is $125. Patients will receive a $10 hospital gift voucher for each urine sample they provide. The total amount that a patient may receive is $50 to $60. At the end of the study, parents who were assigned to the standard advice control group may receive the ETS intervention program without charge, if they so choose. Also, parents in both groups may choose to receive feedback about their child's urine cotinine results at the completion of the study.

ELIGIBILITY:
Inclusion Criteria:

Patient Characteristics

* SJCRH patient with primary diagnosis of any type of cancer.
* ≤17 years of age at the time of enrollment.
* At least one month from diagnosis and in active treatment at the time of enrollment.
* Does not currently use tobacco (defined as abstinence from tobacco during the 30 days preceding the screening assessment as based on patient, 10-17 years of age,and/or parent report).
* Lives with at least one cigarette smoking adult (must be parent or family member/relative) who smokes in their presence (i.e. in the home/hotel, in the same room, in the car, etc) by parent report. Smoking adults will be defined as those who have smoked cigarettes in the past 30 days, per parent report.
* Patient, 10-17 years of age, reads and speaks English.

Parent/Step-Parent/Legal Guardian Characteristics:

* Reads and speaks English.
* Informed consent by institutional guidelines.

Exclusion Criteria:

Patient Characteristics

* Patients with relapse or recurrence of disease within the past month or those with progressive disease.
* Patients in medical crisis as determined by consultation with the child's primary care physician.
* Patients with poor prognosis high-risk malignancies not likely to survive 12 months from diagnosis as documented by child's primary care physician.
* On bone marrow transplant service.

Parent/Step-Parent/Legal Guardian Characteristics:

* Patient's social worker or primary care physician will be consulted prior to parents being approached for enrollment to ensure that the parent is not currently in crisis or distress or have another disabling condition that would preclude participation.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 166 (Actual)
Dates: Start 2002-09; Primary Completion 2010-02 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To determine the efficacy of an Environmental Tobacco Smoke (ETS) exposure intervention compared to a Standard Care Control (SCC) condition, as measured by parent report. | Parent self-reports and patient's urine cotinine levels will be assessed at Baseline, 3, 6, 9, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Sean Phipps, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org